CLINICAL TRIAL: NCT01529892
Title: An Open-Label Study to Evaluate the Impact of Genetic Variation in CYP2D6 on the Pharmacokinetics and Pharmacodynamics of Methamphetamine in Healthy Adults
Brief Title: The Impact of Genetic Variation in CYP2D6 on the Pharmacokinetics and Pharmacodynamics of Methamphetamine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1I
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Methamphetamine Metabolism, CYP2D6 Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methamphetamine EM (Experimental): Extensive metabolizer will be give a single oral 5 mg of duterium labeled methamphetamine
  Interventions: Drug: A single oral 5 mg of duterium labeled methamphetamine
- methamphetamine PM (Experimental): Poor Metabolizers will be give a single oral 5 mg of duterium labeled methamphetamine
  Interventions: Drug: A single oral 5 mg of duterium labeled methamphetamine

INTERVENTIONS:
Drug: A single oral 5 mg of duterium labeled methamphetamine

SUMMARY:
Methamphetamine abuse and addiction are widespread and is causing increasing pressures on social, public health and criminal justice systems worldwide. Some of the risk for developing addiction may be genetic. Identifying specific genotypes and understanding their interactions with the environment may help predict who is at risk for developing a disease. In this study the investigators are evaluating the contribution of differences in one genotype - called CYP2D6 to the removal of methamphetamine from the body. Methamphetamine is removed from the body by special enzymes in the liver. One of these enzymes is called Cytochrome P450 2D6. The activity of 2D6 is genetically determined. Some people have no active 2D6 whereas in others 2D6 is very active. One group of scientists found that people with low 2D6 activity were less likely to become methamphetamine addicts. In this study the investigators will determine the activity of your 2D6 by looking at the CYP2D6 genotype. If low levels of 2D6 decrease the risk of methamphetamine addiction it may be because there is less of the chemicals (called metabolites) made by 2D6. The first step in the metabolism (the process of removal of drugs from the body) of methamphetamine by 2D6 is conversion of methamphetamine to amphetamine and para-hydroxymethamphetamine. 2D6 then converts these to inactive chemicals. In addition to determining your genotype, the investigators are interested in the relationship of genotype with the methamphetamine metabolism. Thus, as part of this study, you will be given a modest oral dose of 5 milligrams of methamphetamine. After receiving the methamphetamine you will need to collect your urine for 24 hours.

The purpose of this study is to investigate the impact of genetic variation in CYP2D6 on the disposition of methamphetamine in the human body as well as its pharmacologic effects to humans.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is healthy, as judged by a responsible physician, with no clinically significant abnormality identified on the laboratory or medical evaluation, including 12-lead ECG, at screening. A subject with a clinical laboratory or laboratory parameter outside the reference range (adjusted for age, if appropriate), may be included only if the Investigator considers that the abnormal finding does not pose additional risk and will not interfere with the study procedures.
2. Male or female, aged 18-55 years inclusive
3. Body weight over 50kg (110 lbs) and body mass index (BMI) of 18.5 to 30 kg/m2 inclusive.
4. Have normal cardiac function including normal blood pressure and heart rate.
5. Have normal renal function as evident by a creatinine clearance >70 ml/min and normal serum creatinine levels
6. The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. A positive urine test for drugs of abuse or alcohol at screening or prior to the start of dosing.
2. Subjects with a clinical history of current alcohol or illicit drug use which, in the opinion of the investigator, would interfere with the subject's ability to comply with the dosing schedule and protocol-specified evaluations.
3. Active Psychiatric disease: DSM-IV diagnosis of a current alcohol, opiate, or sedative hypnotic dependence disorder requiring medical detoxification, history of decompensated schizophrenia, schizophreniform, or schizoaffective disorder; Severe mania, hypomania, agitated behaviour, bipolar disorder or post-traumatic stress disorder within the past 90 days; presence of suicidal behavior two years prior to enrolment or suicidal intent within the past 30 days.
4. The subject has received an investigational drug or participated in any other research trial within 30 days, 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
5. Use of any prescription or non-prescription drugs, vitamins, herbal and dietary supplements within seven days (or 14 days if the drug is a potential CYP2D6 enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study mediation, unless, in the opinion of the Investigator and sponsor, the medication will not interfere with the study procedures or compromise subject safety.
6. Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, intestinal or urinary obstruction, or celiac sprue.
7. History of hypersensitivity to amphetamine-type drugs, or history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
8. Pregnancy or fertile women without adequate means of contraception.
9. Any other medical or psychosocial condition that would preclude useful, safe or consistent participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
urine metabolic ratio | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- St Luke Hospital, Californai Pacific Medical Center, San Francisco, California, United States